CLINICAL TRIAL: NCT01551446
Title: Pilot Assessment of the Effects of Bardoxolone Methyl on Renal Perfusion, Systemic Haemodynamics and Cardiac Function in Patients With Chronic Kidney Disease and Type 2 Diabetes
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: IDMC recommendation for safety concerns
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-1103
Record Dates: First submitted 2012-03-05; First posted 2012-03-12 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — bardoxolone methyl

ARMS (1):
- Bardoxolone Methyl 20mg (Experimental)
  Interventions: Drug: Bardoxolone Methyl

INTERVENTIONS:
Drug: Bardoxolone Methyl — Oral, once daily

SUMMARY:
This study is to evaluate the variability of several pharmacodynamic measures of kidney function, cardiovascular function, cerebral perfusion, and haemodynamics.

ELIGIBILITY:
Inclusion Criteria:

1. Screening eGFR ≥15.0 and ≤60.0 mL/min/1.73 m2;
2. A history of type 2 diabetes; diagnosis should have been made at ≥ 30 years of age (if diabetes developed at a younger age, a fasting C-peptide level must be ≥ 0.1 ng/mL to confirm type 2 diabetes);
3. Male or female patients at least 18 years of age;
4. Treatment with an angiotensin converting enzyme (ACE) inhibitor and/or an angiotensin II receptor blocker (ARB) for at least 6 weeks prior to Study Day 1. The dosage of ACE inhibitor and/or ARB must be stable for 2 weeks prior to and/or during screening (i.e., no change in dosage or medication). Patients not taking an ACE inhibitor and/or ARB, or taking an ACE inhibitor and/or ARB at levels below the goal dose set by K/DOQI guidelines must have a documented medical contraindication (e.g., hyperkalemia, hypotension), which the investigator must provide and discuss with a medical monitor prior to Study Day 1. Patients not taking an ACE inhibitor and/or ARB because of a medical contraindication must have discontinued treatment at least 8 weeks prior to Study Day 1;
5. Mean systolic blood pressure (SBP) ≤160 mmHg and ≥105 mmHg and mean diastolic blood pressure (DBP) ≤90 mmHg during screening; both mean SBP and mean DBP (determined as the average of three readings) must be within the described range during the screening period;
6. Willing to practice methods of birth control (both males who have partners of childbearing potential and females of childbearing potential) during screening, while taking study drug and for at least 30 days after the last dose of study drug is ingested;
7. Serum magnesium level must be ≥1.3 mEq/L (0.65 mmol/L) during the screening period;
8. Willing and able to cooperate with all aspects of the protocol;
9. Willing to and able to give written informed consent for study participation.

Exclusion Criteria:

1. Type 1 diabetes mellitus (juvenile onset). If a history of diabetic ketoacidosis exists, a fasting C-peptide level must confirm type 2 diabetes;
2. Known non-diabetic renal disease (e.g., known polycystic kidney disease, family history of a hereditary form of kidney disease, or congenital absence of one kidney) [nephrosclerosis superimposed on diabetic kidney disease is acceptable];
3. Ongoing clinical investigation with evidence (e.g., unexplained hematuria or red blood cell or white blood cell casts) suggesting non-diabetic renal disease other than nephrosclerosis;
4. History of a renal donation, transplant or a planned transplant from a living donor during the study;
5. Albumin/creatinine (ACR) during screening period greater than 3500 mg/g (395.5 mg/mmol);
6. Hemoglobin A1c level >11.0% (97 mmol/mol) during screening period;
7. Acute dialysis or acute kidney injury within 12 weeks prior to screening or during screening;
8. Clinical signs and/or symptoms of uremia and expected need for renal replacement therapy within 6 weeks following Study Day 1, as assessed by the investigator;
9. Recently active cardiovascular disease defined as:

   * Unstable angina pectoris within 12 weeks before Study Day 1;
   * Myocardial infarction, coronary artery bypass graft surgery, or percutaneous transluminal coronary angioplasty/stent within 12 weeks before Study Day 1;
   * Cerebrovascular accident, including transient ischemic attack within 12 weeks before Study Day 1;
10. Clinical diagnosis of severe obstructive valvular heart disease or severe obstructive hypertrophic cardiomyopathy;
11. Atrioventricular block, 2o or 3o;
12. Administration of a contrast agent that may induce nephropathy within 30 days prior to Study Day 1 or planned during the study;
13. Systemic immunosuppression for more than 2 weeks, cumulatively, within the 12 weeks prior to Study Day 1 or anticipated need for immunosuppression during the study;
14. Total bilirubin, aspartate transaminase (AST), or alanine transaminase (ALT) level greater than the upper limit of normal (ULN) or alkaline phosphatase level >2x ULN on ANY screening laboratory test result;
15. Female patients who are pregnant, intend to become pregnant during the study, or are nursing;
16. BMI < 18.5 kg/m2;
17. Known hypersensitivity to any component of the study drug;
18. Current history of drug or alcohol abuse, as assessed by the investigator;
19. Clinically significant infection requiring intravenous administration of antibiotics or hospitalization within 6 weeks prior to or during the screening period;
20. Hepatitis B surface antigen positive;
21. Diagnosis or treatment of a malignancy in the past 5 years, excluding non-melanoma skin cancer and carcinoma in situ of the cervix, or a condition highly likely to transform into a malignancy during the course of the study;
22. A clinical condition that, in the judgment of the investigator, could potentially pose a health risk to the patient while involved in the study;
23. Participation in a clinical study involving any intervention within 30 days prior to Study Day 1, concurrent participation in such a study, or participation in a prior clinical study involving bardoxolone methyl in any form;
24. Unable to understand verbal or written information in English;
25. Mental incapacity to consent;
26. Contraindications to MRI (implants, pace makers, claustrophobia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2012-11-30 (Actual); Study Completion 2012-11-30 (Actual)

PRIMARY OUTCOMES:
Change in renal perfusion | 20 weeks
  The change in renal perfusion measured by ASL-MRI Scanning

SECONDARY OUTCOMES:
Change in cardiac function | 20 weeks
  The change in cardiac function measured by cardiac MRI scanning
Change in cerebral perfusion | 20 weeks
  The change in cerebral perfusion measured by cerebral ASL MRI
Change in haemodynamic variables | 20 weeks
  The change in the following haemodynamic variables: non-invasive measurement of cardiac output, heart rate, blood pressure and baroreflex sensitivity
Change in arterial stiffness | 20 weeks
  The change in arterial stiffness measured using cartoi-femoral Pulsewave Velocity Assessment and Augmentation Index
Change in body composition | 20 weeks
  The change in body composition measured using Bioelectrical Impedance Analysis
Number of participants with adverse events and serious adverse events | 20 weeks
Plasma concentration of bardoxolone methyl | 20 weeks
Change in cerebral white matter microstructure | 20 weeks
Change in total body water | 20 weeks
  The change in total body water measured using Bioelectrical Impedance Analysis

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/